CLINICAL TRIAL: NCT06431594
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Clinical Activity of GSK5733584 for Injection in Subjects With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Clinical Activity of GSK5733584 for Injection in Participants With Advanced Solid Tumors
Acronym: BEHOLD-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 222730; 2024-513860-25 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors; Neoplasms
Keywords: Solid Tumors; GSK5733584
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants with advanced solid tumors who are refractory or intolerant to established standard therapies
  Interventions: Drug: GSK5733584
- Part 2: Dose Expansion (Experimental): Participants with platinum-resistant ovarian cancer (PROC) and endometrial cancer (EC)
  Interventions: Drug: GSK5733584

INTERVENTIONS:
Drug: GSK5733584 — GSK5733584 will be administered

SUMMARY:
The goal of this study is to assess the safety and tolerability of GSK5733584. The study will also see how the levels of GSK5733584 change over time at different dose amount.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or older (≥18 years).
* Participants with pathologically confirmed advanced solid tumor (who have failed or are intolerant to standard of care).
* PROC cohort

  1. Histologically documented, advanced (metastatic and/or unresectable) high-grade serous/endometrioid ovarian, primary peritoneal, or fallopian tube cancer.
  2. Must have received or are intolerant to 1 but no more than 3 lines of prior systemic therapy.
  3. Platinum-resistant disease, defined as progression or relapse within 6 months after the completion of platinum-based therapy.
  4. Must have had prior bevacizumab if the participant was considered a candidate for this regimen and the regimen is locally available.
  5. Participants with known Folate receptor-α (FR-α) expressing tumors must have received mirvetuximab soravtasine if the participants was considered a candidate for this regimen and the regimen is locally available.
  6. Participants with known Breast cancer susceptibility gene (BRCA) mutated tumors should have received a Poly adenosine diphosphate-ribose polymerase (PARP) inhibitor if the participant was considered a candidate for this regimen and the regimen is locally available.
* Endometrial cancer cohort

  1. Histologically documented, advanced (metastatic and/or unresectable) or recurrent endometrial cancer.
  2. Must have received or are intolerant to 1 but no more than 3 lines of prior systemic therapy.
  3. Must have had prior platinum and PD(L)-1 inhibitor (in same regimen or in separate regimens), if considered a candidate for this regimen and the regimen is locally available.
  4. All epithelial histologies are permitted including carcinosarcoma.
* Participants have at least one target lesion as assessed per the RECIST 1.1
* Tumor tissue from a newly obtained biopsy or archival tumor tissue is required for retrospective detection of B7 homolog 4 (B7-H4) expression by Immunohistochemistry (IHC) in central laboratory and other biomarker analysis. Tissue from a newly obtained biopsy is preferred. If a newly obtained biopsy is not feasible, archival tumor tissue within 2 years prior to the first dose of study drug is acceptable.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 to 2 and no deterioration within 2 weeks before the first dose.
* Have a life expectancy of at least 12 weeks.

Exclusion Criteria:

* Have received any of B7-H4-targeted therapies.
* Have received any of cytotoxic chemotherapy drugs, anti-tumor traditional Chinese medicines or other anti-tumor drugs within 28 days prior to the first dose of study drug; or need to continue these drugs during the study.
* Have received locoregional radiation therapy within 2 weeks prior to the first dose of study drug; more than 30% of bone marrow irradiation or wide-field radiation therapy within 4 weeks prior to the first dose of study treatment.
* Presence of pleural/abdominal effusion/ascites requiring clinical intervention; presence of pericardial effusion
* Major surgery within 28 days prior to the first dose of study treatment.
* Evidence of brain metastasis unless asymptomatic.
* Has inadequate bone marrow reserve or hepatic/renal functions.
* Mean Fridericia-corrected QT interval (QTcF) > 470 millisecond (msec) on resting ECG.
* Evidence of current clinically significant arrhythmias or ECG abnormalities
* Risk factors of prolonged QTc or arrhythmia events,
* Left ventricular ejection fraction (LVEF) < 50%.
* Have severe, uncontrolled or active cardiovascular disorders, serious or poorly controlled hypertension, clinically significant bleeding symptoms or serious arteriovenous thromboembolic events
* Any evidence of current Interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or pneumonitis requiring high-dose systemic glucocorticoids.
* Have received prior therapy with topoisomerase inhibitors or topoisomerase inhibitor Antibody-drug conjugate (ADCs)
* PROC

  1. Primary platinum refractory disease defined as those who have progressed on or within 12 weeks of last dose of first line platinum therapy not permitted.
  2. Non-epithelial carcinoma, clear-cell, mucinous, germ-cell, low-grade serous, or low-grade endometrioid carcinoma not permitted.
* Endometrial cancer a. Mesenchymal tumors of the uterus (uterine sarcomas) not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with dose limiting toxicity (DLT) | Up to 21 days
Part 2: Confirmed Objective Response Rate (ORR) | Up to approximately 28 months
  ORR is defined as the proportion of participants with at least one confirmed Complete Response (CR) or Partial Response (PR) as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

SECONDARY OUTCOMES:
Part 1 and 2: Maximum observed concentration (Cmax) of GSK5733584 and its components: conjugated antibody, total antibody, and small molecule toxin | Up to approximately 31 months
Part 1 and 2: Time to reach Cmax (Tmax) of GSK5733584 and its components: conjugated antibody, total antibody, and small molecule toxin | Up to approximately 31 months
Part 1 and 2: Area under the concentration-time curve (AUC) of GSK5733584 and its components: conjugated antibody, total antibody, and small molecule toxin | Up to approximately 31 months
Part 1: Confirmed Objective Response Rate (ORR) | Up to approximately 31 months
  ORR is defined as the proportion of participants with at least one confirmed CR or PR as defined by RECIST 1.1
Part 1 and 2: Duration of response (DoR) | Up to approximately 31 months
  DoR is defined as the time interval between the date of the first documented response (CR or PR) and the date of the first documented disease progression or death due to any cause
Part 1 and 2: Progression-free survival (PFS) | Up to approximately 31 months
  PFS is defined as the time interval between randomization (or from the first dose of the intervention) and the first documented disease progression or death due to any cause (whichever occurs first).
Part 1 and 2:Number of participants with treatment-emergent Anti-drug antibodies (ADA)/ Neutralizing antibody (NAb) | Up to approximately 31 months
Part 1 and 2: Titers of ADA to GSK5733584 | Up to approximately 31 months
Part 1 and 2: Number of participants with Adverse Events (AEs), and Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) | Up to approximately 31 months
Part 1 and 2: Change from baseline in body temperature (degree Celsius) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in respiratory rate (breaths per minute) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in pulse rate (beats per minute) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in blood pressure [millimetres of mercury (mmHg)] | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in weight [kilogram (kg)] | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in white blood cell count (cells per microliter) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in hemoglobin (grams per deciliter) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from Baseline in Platelet count (cells per microliter) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from Baseline in Red Blood Cell Count (RBC) (million cells per microliter) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from Baseline in haematocrit (Proportion of red blood cells in blood) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from Baseline in Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils (giga cells per litre) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from Baseline in Glucose (fasting), Blood Urea Nitrogen (BUN), Creatinine, Sodium, Potassium, Calcium, Chloride, Magnesium Direct Bilirubin and Total Bilirubin (milligrams per decilitre) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from Baseline in AST/SGOT, ALT/ SGPT, ALP and CPK (International Units per litre) | Baseline (Day -1) and up to approximately 31 months
  Aspartate Aminotransferase (AST) / Serum Glutamic-Oxaloacetic Transaminase (SGOT), Alanine Aminotransferase (ALT)/ Serum Glutamic-Pyruvic Transaminase and (SGPT), Alkaline phosphatase (ALP) and Creatinine Phosphokinase (CPK) will be analysed
Part 1 and 2: Change from baseline in Total Protein and Albumin (Grams per deciliter) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in Amylase and Lipase (Units per liter) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in Estimated glomerular filtration rate (eGFR) (milliliter per minute) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in Prothrombin Time (PT), Partial thromboplastin time (PTT) or Activated Partial Thromboplastin Time (aPTT) (seconds) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in liver panel parameter: International Normalized Ratio (INR) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in routine urine tests: Leukocyte esterase | Baseline (Day -1) and up to approximately 31 months
  Leukocyte esterase measured as negative or positive
Part 1 and 2: Change from baseline in routine urine tests: Occult blood (10^9 Cells Per Liter) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in routine urine tests: potential of hydrogen (pH) value | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in routine urine tests: Protein and bilirubin (Grams Per Liter) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change From Baseline in routine urine tests: Specific Gravity (Ratio) | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in CA-125 tumor marker among ovarian cancer participants [units per milliliter (U/mL)] | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in Thyroid stimulating hormone (TSH) [microunits per milliliter (µU/mL)] | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in free thyroxine (T4) [nanograms per deciliter (ng/dL)] | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in Electrocardiogram (ECG) readings [milliseconds (msec)] | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in Left ventricular ejection fraction (LVEF) [Percentage] | Baseline (Day -1) and up to approximately 31 months
Part 1 and 2: Change from baseline in Eastern Cooperative Oncology Group Performance Scale (ECOG PS) score | Baseline (Day -1) and up to approximately 31 months
  ECOG PS is used for measuring how the disease impacts a patient's daily living abilities. The grades for the scale range from 0 (fully active) to 5 (dead), with increasing severity.
Part 2: Overall Survival (OS) | Up to approximately 31 months
  OS is defined as the time interval between the date of randomization (or from the first dose of the investigational product) and the date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (39):
- United States (8):
  - GSK Investigational Site, Lake Mary, Florida
  - GSK Investigational Site, Fairway, Kansas
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, West Valley City, Utah
- Argentina (3):
  - GSK Investigational Site, Cipoletti Rio Negro
  - GSK Investigational Site, Ciudad de Buenos Aires
  - GSK Investigational Site, Rosario
- Australia (2):
  - GSK Investigational Site, Blacktown, New South Wales
  - GSK Investigational Site, Macquarie University, New South Wales
- GSK Investigational Site, Leuven, Belgium
- Canada (3):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Finland (2):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Tampere
- France (3):
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Villejuif
- Italy (2):
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Rozzano MI
- Japan (3):
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Amsterdam, Netherlands
- South Korea (2):
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
- Sweden (2):
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- United Kingdom (2):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/